CLINICAL TRIAL: NCT01942655
Title: ANRS RF002 Intestipax : Interleukin-23 (IL-23)/Interleukin-12 (IL-12) Imbalance and T Lymphocyte Polarization in HIV Infection
Brief Title: IL-23/IL-12 Imbalance and T Lymphocyte Polarization in HIV Infection
Acronym: INTESTIPAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ANRS RF002 INTESTIPAX
Record Dates: First submitted 2013-08-14; First posted 2013-09-16 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: HIV Reservoirs
Keywords: HIV; Chronic inflammatory bowel disease; Reservoirs; IL-17; IL-23; Intestinal biopsies
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with recto-colic biopsies prescribed (Experimental): 45 patients
  Interventions: Other: Blood sample and recto-colic biopsies

INTERVENTIONS:
Other: Blood sample and recto-colic biopsies

SUMMARY:
Progressive HIV or HIV infection seems to be related to a preferential loss of CD4+ T lymphocytes, especially Th17+, within the mucosal intestinal lymphoid tissue, and with intestinal mucosal damage and bacterial product translocation, which correlates with the hyperactivation of the immune system, therefore with CD4+ T cell loss and prognosis. The objectives of this project are to investigate the correlation between the IL12/IL-23 imbalance and bacterial product translocation, and to study the polarization, infection or depletion of intestinal Th17 ex vivo. The investigators will test the effect of neutralizing anti-IL23 antibodies directed against p40, or less classically, anti- IL-23 p19.

DETAILED DESCRIPTION:
Th17 lymphocytes fight bacterial and fungal intestinal infections. Under combined antiretroviral therapy, even if the plasma viral load is undetectable, hyperactivation can persist, inducing localized replication from reservoirs. In humans, Th17 lymphocyte differentiation and expansion depend on IL-23. The investigators were the first to uncover an imbalance in the respective production of IL-12 and IL-23 in response to Lipopolysaccharide (LPS) in HIV-1 infected patients. IL-23 and its receptor are implicated in the pathogenesis of chronic inflammatory bowel diseases (IBD) like Crohn's disease, where the mucosa is altered by Th17 cells, inducing bacterial product translocation. IBD can be efficiently treated by antibodies directed against Tumor Necrosis Factor-α (TNF-α) or, in current clinical trials, against the p40 chain which is shared by IL-12 and IL-23. Unfortunately, these antibodies inhibit also IL-12. IL-12 is crucial against mycobacteria, which are opportunistic in HIV-infected patients. Antibodies directed against the p19 chain of IL-23 would inhibit Th17 activation more specifically.

The investigators will collect blood and recto-colic biopsies from 15 healthy donors, 15 HIV-infected patients with a viral load higher than 5000 copies/ml and 15 patients with evolutive IBD, to establish a parallel between the two diseases.

The objectives of this project are to study if there is a correlation between the IL12/IL-23 imbalance and bacterial product translocation, and to investigate the polarization, infection or depletion of intestinal Th17 ex vivo. Investigators will test the effect of neutralizing anti-IL23 antibodies directed against p40, or less classically, anti- IL-23 p19.

If these correlations are validated, the investigators will propose anti-IL-23 neutralizing treatment to allow Th17 and intestinal integrity to come back into balance, and therefore to break the vicious cycle of immune system hyperactivation drawn by bacterial translocation.

ELIGIBILITY:
* Age higher than 18
* Able to give written consent
* Recto-colic biopsies prescribed for patient care
* Covered by French Health Insurance System (Social Security) (15 HIV patients with documented detectable HIV viral load in the past 6 months, 15 HIV negative patients with evolutive IBD, 15 HIV negative patients without evolutive IBD)

Exclusion Criteria:

* Absence of coverage by French Health insurance system (Social Security)
* Known progressive malignancy
* Indeterminate colitis
* Known autoimmune diseases other than IBD
* Current chemotherapy or radiotherapy
* Vulnerable populations (children, pregnant women, persons under legal guardianship, or deprived of freedom by judicial or administrative decision)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Multiple measures: IL-17 and IL-23 producing cells in blood, and IL-17 and IL-23 coding mRNA in intestinal biopsies. | 25 months

SECONDARY OUTCOMES:
Multiple measures : number of cells producing IL-23 and Th17 cells in intestinal biopsies | 25 months

OTHER OUTCOMES:
Multiple measures : HIV viral load levels in blood and intestinal biopsies | 25 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigation Clinique BT505, Hôpital Cochin, Paris, France